CLINICAL TRIAL: NCT03473691
Title: Pilot Study of the Antibody-drug Conjugate Glembatumumab Vedotin (CDX-011) Following Doxorubicin (Adriamycin) and Cytoxan as Neo-adjuvant Therapy in Glycoprotein NMB-expressing High Risk Triple Negative Breast Cancer
Brief Title: Pilot Study of Glembatumumab Vedotin Following Doxorubicin and Cytoxan as Neo-adjuvant Therapy in Gp-NMB-expressing High Risk Triple Negative Breast Cancer
Acronym: Breast50
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Pharmaceutical company decided to withdraw funding and not provide drug.
Sponsor: University of Virginia (Other)
Collaborators: Celldex Therapeutics (Industry)
Responsible Party: Principal Investigator, Patrick Dillon, MD, Principal Investigator, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TBDBreast50
Record Dates: First submitted 2018-02-14; First posted 2018-03-22 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — glembatumumab vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Glembatumumab vedotin (GV) (Experimental)
  Interventions: Drug: Glembatumumab Vedotin

INTERVENTIONS:
Drug: Glembatumumab Vedotin — Standard neo-adjuvant dose-dense doxorubicin 60 mg/m2 and Cytoxan 600 mg/m2 IV every 14 days for 4 cycles followed by GV 1.9 mg/kg IV every 21 days for 4 cycles.
  Other Names: CDX-011

SUMMARY:
This is a single arm, pilot study assessing safety/feasibility and efficacy of neo-adjuvant glembatumumab vedotin (GV) in patients with high risk triple negative breast cancer (TNBC) with glycoprotein-NMB (gpNMB) expression ≥ 25%. Primary endpoints will be safety/feasibility, and secondary endpoints will be rates of pathologic complete response (pCR), and measurements of growth differentiation factor-11 (GDF11) and glycoprotein NMB (gpNMB) expression.

DETAILED DESCRIPTION:
Patients will receive neo-adjuvant dose-dense (DD) doxorubicin (Adriamycin)/cyclophosphamide (AC) followed by GV. After completion of neo-adjuvant therapy, all patients will undergo lumpectomy (with radiation therapy) or mastectomy, and tissue will be assessed for residual disease to determine rates of pCR. Tumor tissue will be obtained by core needle biopsy and at the time of surgery for use in the correlative studies.

ELIGIBILITY:
Inclusion Criteria:

1. Willingness and ability to provide written informed consent and to comply with the study protocol as judged by the investigator.
2. Patients diagnosed with triple negative breast cancer, (stages II-III, or high risk T1c disease) found to have gpNMB expression at or above 25%), and who are appropriate candidates for neo-adjuvant therapy. Patients must be willing to undergo lumpectomy (with radiation therapy) or mastectomy following neo-adjuvant therapy.
3. Subjects may be female or male.
4. ECOG Performance Status of 0-2.
5. Age ≥ 18 years.
6. Subject must have a life expectancy ≥ 6 months.
7. Absolute neutrophil count ≥ 1,500 cells/mm3
8. Platelets ≥ 100,000 cells/mm3
9. Hemoglobin ≥ 9g/dl (Note: The use of transfusion to achieve Hemoglobin ≥ 9 g/dl is acceptable)
10. Serum creatinine OR GFR ≤ 1.5 x institutional upper limit normal (IULN)
11. Bilirubin ≤ 1.5 x IULN OR Direct Bilirubin ≤ULN for patients with total bilirubin levels >1.5×ULN
12. ALT and AST ≤ 2.5 IULN
13. Alkaline phosphatase ≤ 2.5 IULN
14. Women of childbearing potential (WOCBP) and men must agree to use adequate contraception prior to study entry and for at least 1 year following last dose of study drug.

    a. WOCBP includes any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation or bilateral oophorectomy) or is not postmenopausal [defined as amenorrhea ≥ 12 consecutive months; or women on hormone replacement therapy with documented serum follicle stimulating hormone (FSH) level > 35 mIU/mL]

    i. Prior to study enrollment, WOCBP must be advised of the importance of avoiding pregnancy during trial participation and for at least 1 year following participation and the potential risk factors for an unintentional pregnancy

ii. The following birth control methods are allowed during the study: Barrier methods (Intra-uterine device (IUD), Diaphragm with spermicide, Cervical cap with spermicide, Condom with spermicide) or Abstinence (no heterosexual activity)

b. Non-vasectomized males must agree to use adequate contraception for at least 120 days after the last dose of study drug

i.The following birth control methods are allowed during the study: Partner is not WOCBP or is taking hormonal contraceptives, Barrier methods (Intra-uterine device (IUD), Diaphragm with spermicide, Cervical cap with spermicide, Condom with spermicide) or Abstinence (no heterosexual activity)

ii. Males must also abstain from sperm donations for at least 120 days after the last dose of study drug

Exclusion Criteria:

1. Patients that have received more than one cycle of neo-adjuvant doxorubicin and cyclophosphamide prior to enrolling on the study.*
2. Prior radiation therapy for this breast cancer. Prior radiation for other malignancy must have been completed >12 weeks prior to on-study date.
3. Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 3 years; non-invasive conditions such as carcinoma in situ of the breast, oral cavity, or cervix are all permissible.
4. Subjects who are receiving any investigational agents or have had any investigational agent within the 30 days prior to on-study date
5. Subjects who are unable or unwilling to discontinue use of prohibited medications including long-term use of systemic corticosteroids (equivalent to ≥ 10 mg prednisone for ≥1 month within 1 month of study enrollment).
6. Subject is unable or unwilling to participate in a study related procedure
7. Pregnant and breastfeeding women. See Pre-Study Assessments section for more information on pregnancy tests.
8. Subject is a prisoner
9. Subjects with known acute hepatitis, human immunodeficiency virus (HIV) or active infections that require parenteral antibiotics.
10. Significant history of uncontrolled cardiac disease defined as uncontrolled hypertension, unstable angina, or myocardial infarction within the last 4 months, and uncontrolled congestive heart failure.
11. A serious uncontrolled medical disorder that in the opinion of the Investigator would impair the ability of the subject to receive protocol therapy.
12. Subjects with history of or evidence upon physical examination of central nervous system disease including primary brain tumor, seizures not controlled with standard medical therapy, any brain metastases, or history of cerebrovascular accident (CVA, stroke), transient ischemic attack (TIA), or subarachnoid hemorrhage within six months of study entry.
13. Baseline neuropathy > grade 2
14. Subjects with a known history of immunogenic response or allergic reactions attributed to compounds of similar chemical composition to dolastatin or auristatin
15. Abnormal cardiac function, defined as a left ventricular ejection fraction (LVEF) < 50% by echocardiogram (ECHO) or multigated acquisition scan (MUGA) * If a patient has undergone one cycle of chemotherapy, he or she must have recovered from all adverse events to ≤ grade 1 to meet the above inclusion criteria. Labs collected prior to initiation of AC treatment may be used for eligibility, as long as they are collected in the required 28 day window. Patients that have received one cycle of AC prior to enrollment will receive 3 additional cycles of AC to complete a total of 4 cycles prior to starting GV.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-05-01 (Estimated); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) | Adverse events will be assessed from the time of consent through 30 days after participants complete GV treatment (unless study treatment is stopped for safety or investigator or participant decision, study treatment will last 25-28 weeks)
  Adverse events will be assessed using the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03
Proportion of patients who complete the 4 cycles of GV within 15 weeks of the first dose of GV (without dose limiting adverse events). | Within 4 months of the last patient enrollment
  To assess feasibility, the proportion of patients who receive the intended dose within 15 weeks of the first dose will be estimated with an 80% confidence interval.
Number of discontinuations due to AEs | During each participant's study treatment. Unless study treatment is stopped for safety or investigator or participant decision, study treatment will last about 22 weeks.
  Adverse events will be assessed using the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03. Participants that discontinue study treatment because of AEs based on protocol-defined stopping rules will be included.

SECONDARY OUTCOMES:
Efficacy | 3-6 weeks after last GV infusion for each patient
  Rates of pathologic complete response (pCR) following GV therapy
Growth Differentiation Factor-11 (GDF11) expression in the tumor | Prior to therapy (in the 28 days prior to starting study treatment) and 3-6 weeks after last GV infusion for each patient.
  GDF11 expression by immunohistochemistry prior to and following doxorubicin/cyclophosphamide and GV therapy
Glycoprotein-NMB (gpNMB) expression in the tumor | Prior to therapy (in the 28 days prior to starting study treatment) and 3-6 weeks after last GV infusion for each patient
  gpNMB expression by immunohistochemistry prior to and following doxorubicin/cyclophosphamide and GV therapy

OTHER OUTCOMES:
Peripheral circulating CD8 and CD4 T cell ratio | Prior to therapy (in the 28 days prior to starting study treatment) and at the last treatment with GV (about 22 weeks after starting study treatment).
  Blood will be collected in order to assess the proportions of CD8 and CD4 t cells.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Dillon, MD, Principal Investigator — University of Virginia